CLINICAL TRIAL: NCT05053789
Title: Efficacy of Different Treatment Regimens With Chitosan-N- Acetylcysteine (Lacrimera®) in Moderate-to-severe Dry Eye Disease: A Pilot Study
Brief Title: Efficacy of Different Treatment Regimens With Chitosan-N- Acetylcysteine in Moderate-to-severe Dry Eye Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Medical device expired
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Lacrimera Efficacy
Record Dates: First submitted 2021-09-01; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Eye Diseases
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The study will be carried out in an observer-masked fashion, therefore the investigator performing the measurements will not be informed about the treatment group that patients are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): After enrolment into the study and randomization to the study group (V0) and baseline examinations (V1), patients will receive 1 drop of Lacrimera at the study site and will be instructed to apply one drop of C-NAC into both eyes before bedtime for the following 5 consecutive days and return for a follow-up visit after 7±1 days (V2). Patients will complete a diary describing symptoms during the day, use of Lacrimera and potential side effects until the next visit. If the NEI grading is ≤1 OR the OSDI score <20 at the next visit, treatment with Lacrimera will be discontinued and one further physical follow-up appointment will be arranged, which will take place 28±2 days after the last physical visit.
  Interventions: Device: Lacrimera
- Group 2 (Active Comparator): The study days are conducted in the same way as for the study group. Patients of the control group will receive preservative-free, Hyaluronic-acid containing eyedrops (Hylo-Vision® sine) for 4 times a day as control.
  Interventions: Device: Hylo-Vision

INTERVENTIONS:
Device: Lacrimera — A new preservative-free formulation of eye drops consists of a novel biopolymer, chitosan-N-acetylcysteine (C-NAC; Lacrimera®, Croma-Pharma GmbH, Leobendorf, Austria), which electrostatically binds to the mucine layer of the tear film forming a glycocalyx-like structure.
  Arms: Group 1
Device: Hylo-Vision — Preservative-free, Hyaluronic-acid containing eyedrops (Hylo-Vision® sine).
  Arms: Group 2

SUMMARY:
Aim of this pilot study is to evaluate the best treatment regime of Chitosan-N-Acetylcysteine (Lacrimera®) compared to preservative-free, Hyaluronic-acid containing eyedrops (Hylo-Vision® sine).

DETAILED DESCRIPTION:
The present pilot study seeks to investigate the best fitting treatment regime of moderate-to-severe DED with C-NAC compared to preservative-free, Hyaluronic-acid containing eyedrops (Hylo-Vision® sine) by applying a randomized, prospective, adaptive, controlled design.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 22 years
* Corneal staining (marked to severe; NEI grading scale >=10)

Exclusion Criteria:

* Usage of eye drops other than lubricants (e.g. antibiotics, steroids, cyclosporin-A)
* Usage of systemic antibiotic therapy
* Any pathology of the ocular surface except dry eye disease (e.g. corneal scarring, cornea ectasia)
* Ocular surgery within prior 3 months to screening
* Preceding refractive corneal surgery (e.g. LASIK)
* Ocular injury within prior 3 months
* Ocular herpes of eye or eyelid within prior 3 months
* Active ocular infection
* Active ocular inflammation or history of chronic, recurrent ocular inflammation within prior 3 months
* Eyelid abnormalities that affect lid function
* Ocular surface abnormality that may compromise corneal integrity
* Pregnancy and nursing women (in women of childbearing age a pregnancy test will be performed before inclusion into the study)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Duration of treatment | 1 month
  Duration of treatment in days until objectively confirmed recovery (NEI (National Eye Institute) grading ≤1 OR OSDI (Ocular Surface Disease Index) score <20, either 7±1, 14±1, 21±1 or 28±1 days) in the study group compared to the control group.

SECONDARY OUTCOMES:
Change in BUT (Break Up Time) | 1 month
  Change in BUT (Break Up Time) at different visits in both groups. Fluorescein Break Up time is measured after instillation of 100 μl fluorescein into the inferior fornix. Using a stopwatch time after the last blink until the first break up of the tear film is recorded. Three consecutive measurements are performed, and the average is calculated.
  Non-invasive first and averaged BUT is measured three times and averaged afterwards using the Dry eye module build into the corneal tomography device (Sirius, CSO, Italy).
Change in NI-BUT (Non-invasive Break Up Time) | 1 month
  Change in NI-BUT (Non-invasive Break Up Time) at different visits in both groups. The Sirius device is a routinely used device for the detailed assessment of the cornea and the tear film. NI-BUT is assessed by monitoring placido discs (Sirius, CSO, Italy) projected onto the cornea. 3 consecutive measurements are made in every eye.
OSDI (Ocular Surface Disease Index) | 1 month
  OSDI (Ocular Surface Disease Index) at different visits in both groups. The OSDI Questionnaire is a standardized questionnaire to evaluate the subjective disease burden caused by dry eye syndrome. The patients answer up to 12 questions regarding their symptoms. Thereafter, the OSDI Score is calculated.
Flourescein staining / Lissamin green staining grading using the NEI Score (National Eye Institute) | 1 month
  Lissamin green staining at different visits in both groups using the NEI Score. Fluorescein and Lissamin green dye will be used to examine the anterior surface of the human eye. Anterior Segment Photography will be used to document the findings, which are graded using the National Eye Institute (NEI) grading scale.
Change in number of MMP-positive eyes (Matrix Metallopeptidase 9) | 1 month
  Change in number of MMP-positive eyes in both groups (Matrix Metallopeptidase 9). MMP-9 is an inflammatory marker of the ocular surface. InflammaDry® allows to indicate elevated levels of MMP-9 in tear fluid by microfiltration technology. Patients will be instructed to look upward, and the lower eye lid will be pulled downward gently. Samples will be collected by dabbing a tear sample collector in 6-8 locations on the palpebral conjunctiva. The test is routinely performed in our dry eye unit.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, PrimUnivPrDr, Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- Vienna Institute for Research in Ocular Surgery, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No